CLINICAL TRIAL: NCT03244241
Title: Basal-bolus Insulin Therapy With Insulin Degludec and Insulin Aspart Versus Standard Therapy for the Inpatient Management of Type 2 Diabetes: the IDA2 Study
Brief Title: Basal-bolus Insulin Therapy Versus Standard Therapy for the Inpatient Management of Type 2 Diabetes: the IDA2 Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Merete Bechmann Christensen (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor-Investigator, Merete Bechmann Christensen, Principle investigator, Hvidovre University Hospital
Organization: Hvidovre University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1177-2744
Record Dates: First submitted 2017-06-07; First posted 2017-08-09 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes, inpatient diabetes management, basal-bolus insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin degludec

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator): Basal-bolus insulin regime with Insulin Degludec and insulin aspart
  Interventions: Drug: Insulin Degludec 100 UNT/ML [Tresiba]
- Standard (No Intervention): Standard treatment according to hospital guidelines with sliding scale insulin

INTERVENTIONS:
Drug: Insulin Degludec 100 UNT/ML [Tresiba] — Basal-bolus insulin regime
  Arms: Intervention

SUMMARY:
Hyperglycemia during admission is associated with increased rate of complications and longer hospital stays, thus insulin treatment is recommended for all diabetes patients with hyperglycemia. Inpatient studies of non-critically ill patients show better glycemic control with the use of basal-bolus insulin therapy compared to sliding scale insulin therapy, but increased rates of hypoglycemia. The investigators hypothesize that basal-bolus insulin therapy with a new ultra-long-action basal insulin can treat hyperglycemia more efficiently than sliding scale insulin, with few episodes of hypoglycemia.

DETAILED DESCRIPTION:
The aim of this study is to investigate and compare the efficacy and safety of basal-bolus insulin therapy using the insulin analogue, insulin degludec once daily and insulin aspart before meals versus standard therapy with sliding scale insulin in non-critical ill hospitalized patients with type 2 diabetes.

The design of the trial is an open, randomized controlled trial with two parallel arms (treatment arm and control arm). Randomization is 1:1.

ELIGIBILITY:
Inclusion Criteria:

* History of type 2 diabetes for at least 6 months
* Age 18 - 90 years
* Pre-meal plasma glucose in the range 10 - 22,2 mmol/L prior to inclusion
* Expected hospital stay longer than 4 days

Exclusion Criteria:

* Hyperglycemia without known history of type 2 diabetes
* Type 1 diabetes mellitus
* Severely impaired renal function (eGFR ≤ 30 mL/min/1,73 m2)
* Severe hepatic disease
* Cardiac disease defined as: Decompensated heart failure (NYHA class III-IV) and/or diagnosis of unstable angina pectoris and/or myocardial infarction within the last 6 months
* Pregnant or lactating women or fertile female patients not using chemical, hormonal or mechanical contraceptives or not in menopause (i.e. must not have had regular menstrual bleeding for at least one year)
* Planned treatment during hospital stay with intravenous glucose/ insulin for ≥ 12 hours
* Treatment at admission or planned treatment during hospital stay with parenteral nutrition or enteral nutrition (i.e. gastroenteric tube feeding)
* Treatment at admission or planned treatment during hospital stay with high dose glucocorticoids (>40 mg)
* History or presence of malignancy (except basal skin cancer) unless a disease-free period exceeding five years
* Presence of alcohol or drug abuse
* Inability to understand the written information or incapability to provide informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-04-01 (Estimated); Study Completion 2018-04-01 (Estimated)

PRIMARY OUTCOMES:
Difference in mean daily plasma glucose between the two groups | Duration of hospital stay, an expected average of 8 days
  Difference in mean daily plasma glucose between the two groups, calculated by using the four daily pre-meal and bedside PG values per patient.

SECONDARY OUTCOMES:
Mean number and rates of hypoglycemic events (PG ≤ 3.9 mmol/L) | Duration of hospital stay, an expected average of 8 days
  Based on bedside PG measures and on CGM data
Time spent in glycemic range | Duration of hospital stay, an expected average of 8 days
  Based on bedside PG measures and on CGM data
Time spent in hyperglycemic range | Duration of hospital stay, an expected average of 8 days
  Based on bedside PG measures and on CGM data
Length of hospital stay | Duration of hospital stay, an expected average of 8 days
  Mean duration of hospital stay
Difference in insulin dose between groups | Duration of hospital stay, an expected average of 8 days
  Calculated as mean insulin dose during admission
Number of hospital acquired infections during admission | Duration of hospital stay, an expected average of 8 days
  Data from hospital record
Number of post-discharge infections or re-admissions 1 month after discharge | 1 month
  Data collected on follow-up 1 month after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten B Norgaard, DMSC, Principal Investigator — Hvidovre University Hospital
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Undecided